CLINICAL TRIAL: NCT02699034
Title: Cardiovascular Magnetic Resonance-Guided Radiofrequency-Ablation for Atrial Flutter: Evaluation of a Tailored Interventional Guidance and Tracking System
Brief Title: Cardiovascular Magnetic Resonance-Guided Radiofrequency-Ablation for Atrial Flutter
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recommendation by BfArM after interim analysis
Sponsor: University of Leipzig (Other)
Collaborators: Heart Center Leipzig - University Hospital (Other); Philips Healthcare (Industry); Imricor Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-IMR
Record Dates: First submitted 2016-02-19; First posted 2016-03-04 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Atrial Flutter
Keywords: real-time MRI; electrophysiology study; atrial flutter ablation; active tracking
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ablation for typical atrial flutter (Experimental): This group receives an MR-guide ablation for atrial flutter with the study device ( Vision-MR ablation catheter )
  Interventions: Procedure: ablation for typical atrial flutter; Device: Vision-MR ablation catheter

INTERVENTIONS:
Procedure: ablation for typical atrial flutter
Device: Vision-MR ablation catheter

SUMMARY:
The purpose of this clinical study is to evaluate the and performance of the Imricor Medical Systems, Inc. (Imricor) MR Ablation Catheter when used with related accessories for the treatment of type I atrial flutter. The Vision Ablation Catheter and its accessories have been designed for use under fluoroscopic or magnetic resonance guidance. The study will be a single center study conducted at the Leipzig University Hospital Heart Center in Germany. The study population will consist of adult patients requiring ablation for type I atrial flutter.

DETAILED DESCRIPTION:
The study will be a single center study conducted at the Leipzig University Hospital Heart Center in Germany. 35 subjects including 5 roll-in subjects meeting inclusion/exclusion criteria will participate in the study. This study requires the use of investigational products from two independent manufacturers: Imricor and Philips. Imricor has developed the ablation catheter with related accessory cables and electrophysiology (EP) recorder/stimulator system. Philips has developed an image guidance and mapping system that is compatible with the Imricor products.

The Vision-MR Ablation Catheter will be used in conjunction with the following investigational products: Advantage-MR EP Recorder/Stimulator, Vision-MR Ablation Cable Set, Vision-MR Diagnostic Cable, the interventional MRI Suite (iSuite) image guidance and mapping system, and a dStream Interface (dSIF-FE). With the exception of iSuite and dSIF-FE, which are manufactured by Philips, Imricor will provide all investigational devices used in the study.

Each procedure will require two single-use Vision-MR Ablation Catheters and one each of the two single-use accessory catheter cables.

Ablation for the treatment of arrhythmia is an inherently complex procedure. Use of the investigational products listed above under MR guidance is an emerging approach to performing the interventional electrophysiology procedure.

The study population will consist of adult patients requiring ablation for type I atrial flutter.

Study subjects will require a follow-up visit or telephone call at seven days post procedure. Accordingly, the expected total study duration is approximately 9 months with study start planned for March 2016.

ELIGIBILITY:
Inclusion Criteria:

* First time indication for ablation for type I atrial flutter.
* Patients willing and able (mentally and physically capable per physician's discretion) to understand the investigational nature, potential risks and benefits of the study and able to provide written informed consent to participate in the study and agree to comply with follow-up visits and evaluation
* Patients able to receive anticoagulation therapy to achieve adequate anticoagulation

Exclusion Criteria:

* Contraindication for MRI diagnostic exam
* A cardiac ablation or cardiac surgery within 180 days prior to enrollment
* Documented intracardiac thrombus, tumor, bleeding, clotting or other abnormality that precludes catheter introduction and placement
* Myocardial infarction within 60 days prior to enrollment
* Current unstable angina
* History of cerebrovascular event (within 180 days prior to enrollment)
* Patients with an ejection fraction less than or equal to 35% within 90 day prior to enrollment
* Permanent leads in or through the right atrium
* Clinically significant structural heart disease (including tricuspid valve regurgitation, tricuspid valve stenosis or other congenital heart disease) that would preclude catheter introduction and placement, as determined by the Investigator
* Uncompensated congestive heart failure (NYHA Class III or IV)
* Arrhythmia is secondary to electrolyte imbalance, thyroid disease, or other reversible or non-cardiovascular cause
* Known sensitivity to heparin or warfarin
* Active or systemic infection
* Any other significant uncontrolled or unstable medical condition (including but not limited to hypertension and diabetes)
* contraindication for conventional ablation procedure know allergy against radiocontrast agents renal insufficiency with glomerular filtration rate < 30ml/min/1,73m2
* Women who are pregnant or plan to become pregnant within the course of their participation in the investigation or who are breastfeeding
* Life expectancy of less than 12 months
* Patients with prosthetic valves
* Contraindicated for transfemoral venous access
* Older than 75 years
* Current enrollment in any other clinical investigation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06-05 (Actual); Study Completion 2016-10-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with bidirectional cavo-tricuspid isthmus block after intervention | 9 months
  Acute success defined as the demonstration of the established electrophysiological endpoint (e.g. bidirectional cavo-tricuspid isthmus block after radiofrequency application in the cavo-tricuspid isthmus) with the investigational device. Historically, the acute success rate for RF ablation of type I atrial flutter is 72%. Analysis will be based on a binomial proportion and expressed as a percentage. For a total of N subjects with S achieving success, the percentage, represented as P, will be calculated as P = 100*S/N.
Incidence of Treatment-Emergent Serious Adverse Events [Safety]) | 9 months
  The primary safety endpoint is the rate of serious adverse events (SAEs) related to the device or procedure. Analysis will be based on a binomial proportion and expressed as a percentage. For a total of N subjects with S experiencing an SAE related to the device or procedure, the percentage, represented as P, will be calculated as P = 100*S/N.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Hindricks, MD, Principal Investigator — Heart Center Leipzig
Locations (1):
- Heart Center Leipzig, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hilbert S, Sommer P, Gutberlet M, Gaspar T, Foldyna B, Piorkowski C, Weiss S, Lloyd T, Schnackenburg B, Krueger S, Fleiter C, Paetsch I, Jahnke C, Hindricks G, Grothoff M. Real-time magnetic resonance-guided ablation of typical right atrial flutter using a combination of active catheter tracking and passive catheter visualization in man: initial results from a consecutive patient series. Europace. 2016 Apr;18(4):572-7. doi: 10.1093/europace/euv249. Epub 2015 Aug 27. PMID 26316146
- See also: Imricor website — http://www.imricor.com